CLINICAL TRIAL: NCT01202409
Title: Phase II Study of Panitumumab in KRAS Wild-type Locally Advanced or Metastatic Adenocarcinoma of the Small Bowel or Ampulla of Vater
Brief Title: CAPOX in KRAS Wild-Type Advanced Adenocarcinoma of the Small Bowel or Ampulla of Vater
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0458; NCI-2012-01894 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Gastrointestinal Cancer
Keywords: Ampulla of Vater; Adenocarcinoma of the small bowel; Metastatic; Kirsten rat sarcoma; KRAS; Capecitabine; Xeloda; Oxaliplatin; Eloxatin; CAPOX; Panitumumab; Vectibix
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasm Metastasis | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panitumumab (Experimental): Starting Dose of Panitumumab: 9 mg/kg by vein over 60 minutes on day 1 of a 14 day cycle.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Starting Dose Level: 9 mg/kg by vein over 60 minutes on day 1 of a 14 day cycle.
  Other Names: Vectibix

SUMMARY:
The goal of this clinical research study is to learn if panitumumab can help to control advanced cancer of the small bowel or ampulla of Vater. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Panitumumab is designed to "turn off" a protein that is important in cell growth. This may stop the growth of cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive the study drug during 14 day study "cycles."

On Day 1 of every cycle, you will receive panitumumab by vein over about 60-90 minutes.

Study Visits:

On or before Day 1 of each cycle:

* You will have a physical exam, including measurement of your weight.
* Your performance status will be recorded.
* You will be asked about any symptoms you may be experiencing and any drugs you may be taking.
* Blood (about 2 tablespoons) will be drawn for routine tests.

Every 4 cycles:

* You will have a chest X-ray or a computed tomography (CT) scan of your chest to check the status of the disease.
* You will have a CT or MRI scan to check the status of the disease. If your scan shows that you are responding to the treatment, you will have another CT or MRI scan 6 weeks later.

Length of Study:

You may continue receiving the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

End-of-Treatment:

After you stop taking the study drugs for any reason, you will have an end-of-treatment visit. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight.
* Your performance status will be recorded.
* You will be asked about any symptoms you may be experiencing and any drugs you may be taking.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a CT or MRI scan of the abdomen and pelvis to check the status of the disease.

Follow-Up:

Thirty (30) days after your last dose of study drug(s), you will be asked about any symptoms you may be experiencing and any drugs you may be taking. If you are unable to come to MD Anderson for this, the study staff will call you and ask you these questions. This call will last about 30 minutes.

You will then be called every 3 months and asked the same questions. Each call will last about 15-30 minutes.

If you are taken off study treatment for reasons other than the disease getting worse, you will have a CT or MRI scan of the abdomen and pelvis to check the status of the disease every 12 weeks (+/- 2 weeks) after the End-of-Treatment visit. This will be done until the disease gets worse and if you do not start any other anti-cancer treatment.

This is an investigational study. Panitumumab is commercially available and FDA approved to treat a certain type of colorectal cancer. Its use in this type of cancer is investigational.

Up to 27 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed adenocarcinoma of the small bowel or ampulla of Vater that is either unresectable or metastatic.
2. Adequate tumor tissue available for KRAS mutational analysis or known KRAS wild-type status.
3. Prior progression on or intolerance to treatment with a fluoropyrimidine and oxaliplatin. Recurrence of disease within 6 months from the completion of adjuvant therapy with both a fluoropyrimidine and oxaliplatin is considered progression.
4. Patients must have measurable disease as per the revised Response Evaluation Criteria In Solid Tumors (RECIST) criteria (Version 1.1).
5. If radiation was previously received, the measurable disease must be outside the previous radiation field, unless this area has demonstrated evidence of radiographic growth.
6. A minimum of 2 weeks must have elapsed from completion of any prior chemotherapy or radiotherapy or surgery and the start date of study therapy.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 2.
8. Adequate organ function including: a) Absolute neutrophil count (ANC) =/>1,000/ul; b) Platelets =/>75,000/ul; c) Total bilirubin =/< 1.5 x ULN; in patients with known Gilbert's syndrome direct bilirubin =/<1.5 x ULN will be used as organ function criteria, instead of total bilirubin; d) AST (SGOT)/ALT (SGPT) < 3 x ULN; e) Creatinine <2 x ULN.
9. Negative urine or serum pregnancy test in women with childbearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization), within one week prior to initiation of treatment.
10. The effects of panitumumab on the developing fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation, and for six months following the completion of therapy. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately.
11. Patients must sign an Informed Consent and Authorization indicating that they are aware of the investigational nature of this study and the known risks involved.
12. Magnesium level =/> lower limit of normal.

Exclusion Criteria:

1. Prior anti-epidermal growth factor receptor antibody therapy (eg. panitumumab or cetuximab) or prior small molecule anti-epidermal growth factor receptor therapy (eg. erlotinib) for adenocarcinoma of the small bowel or ampulla of Vater.
2. Patients may not be receiving any other investigational agents nor have received any investigational drug 30 days prior to enrollment.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit adherence with study requirements.
4. Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.
5. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with panitumumab, breast feeding must be discontinued.
6. Age <18 years. Because no dosing or adverse event data are currently available on the use of panitumumab in patients <18 years of age, children are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11-02 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Overman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gulhati P, Raghav K, Shroff R, Varadhachary G, Javle M, Qiao W, Wang H, Morris J, Wolff R, Overman MJ. Phase II Study of Panitumumab in RAS Wild-Type Metastatic Adenocarcinoma of Small Bowel or Ampulla of Vater. Oncologist. 2018 Mar;23(3):277-e26. doi: 10.1634/theoncologist.2017-0568. Epub 2017 Dec 19. PMID 29259073
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine + Panitumumab + Oxaliplatin: Capecitabine 750mg/m2 oral twice daily, Days 1 - 14 and Panitumumab 9 mg/kg IV over 60 minutes on Day 1 and Oxaliplatin 130 mg/m2 IV over 2 hours Day 1 of 21-day cycle.
Period: Overall Study
Arm/Group | Capecitabine + Panitumumab + Oxaliplatin
Started | 19
Completed | 11
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Ineligible - KRAS mutants | 7

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine + Panitumumab + Oxaliplatin
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 60 [39 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 100 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine + Panitumumab + Oxaliplatin
Number analyzed (Participants) | 19
Participants | 19

2. Secondary Outcome: Overall Progression-free Survival (PFS) for CAPOX and Panitumumab
Description: Time interval in months from date of first treatment until the date of first documented progression of participants.
Time Frame: 7.6 months
Measure: Median (Full Range); unit: months
Arm/Group | Capecitabine + Panitumumab + Oxaliplatin
Number analyzed (Participants) | 13
months | 2.4 [1 to 7.6]

ADVERSE EVENTS:
Time Frame: Adverse event collection from date of first treatment to 8 years
Arm/Group | Capecitabine + Panitumumab + Oxaliplatin
All-Cause Mortality (participants affected / at risk) | 19/19
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Panitumumab + Oxaliplatin (N=19)
Skin Infection (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Panitumumab + Oxaliplatin (N=19)
Abdominal pain (Gastrointestinal disorders) | 2
Alanine Aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 3
Anemia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dry Eye (Eye disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Eye disorders - other (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nail infection (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral hemorrhage (Gastrointestinal disorders) | 1
Palmmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Paronychia (Skin and subcutaneous tissue disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 11
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Respiratory, Thoracic and Mediastinal Disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disoreders - Other (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT01202409/Prot_SAP_000.pdf